CLINICAL TRIAL: NCT03233555
Title: Extended Cancer Education for Longer-Term Survivors (EXCELS) In Primary Care
Brief Title: Extended Cancer Education for Longer-Term Survivors in Primary Care for Patients With Stage I-II Breast or Prostate Cancer or Stage I-III Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 131318; NCI-2017-01185 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2013003309; 131318 (Other: Rutgers Cancer Institute of New Jersey); R01CA176838 (NIH)
Record Dates: First submitted 2017-07-19; First posted 2017-07-28 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Stage I Breast Cancer; Stage I Colorectal Cancer AJCC v6 and v7; Stage I Prostate Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage II Colorectal Cancer AJCC v7; Stage II Prostate Cancer; Stage IIA Breast Cancer; Stage IIA Colorectal Cancer AJCC v7; Stage IIA Prostate Cancer; Stage IIB Breast Cancer; Stage IIB Colorectal Cancer AJCC v7; Stage IIB Prostate Cancer; Stage IIC Colorectal Cancer AJCC v7; Stage III Colorectal Cancer AJCC v7; Stage IIIA Colorectal Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (brochure) (Active Comparator): Participants receive National Cancer Institute's Facing Forward brochure.
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (EXCELS website) (Experimental): Participants have untimed access to the EXCELS mobile web application.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (Healthcare coaching call) (Experimental): Participants also receive 4 quarterly calls of 15-20 minutes each over 3 months. These calls focus on checking if patients have received preventive and cancer related follow-up care.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention
- Arm IV (EXCELS website, health coaching calls) (Experimental): Participants have access to EXCELS as in Arm II. Participants also receive 4 calls as in Arm III.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Informational Intervention — Receive brochure
  Arms: Arm I (brochure)
Other: Internet-Based Intervention — Have access to EXCELS
  Arms: Arm II (EXCELS website); Arm IV (EXCELS website, health coaching calls)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive quarterly calls
  Arms: Arm III (Healthcare coaching call); Arm IV (EXCELS website, health coaching calls)

SUMMARY:
This study tests four different methods of educating patients about follow-up care (NCI facing forward, brochure, EXCELS website alone, EXCELS health coaching alone and EXCELS website & health coaching combination) after cancer treatment ends. While it is known that patients need information to guide follow-up it remains unknown how to best provide this in primary care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop the EXCELS intervention to facilitate engaged self-management of cancer follow-up for cancer survivors.

II. Evaluate the efficacy of EXCELS intervention in a small randomized controlled trial.

III. Assess/refine intervention usability and acceptability for primary care patients.

OUTLINE:

PHASE I: EXCELS intervention is developed and assessed.

PHASE II: Participants are randomized into 1 of 4 arms.

ARM I: Participants receive National Cancer Institute's Facing Forward brochure.

ARM II: Participants have untimed access to the EXCELS mobile web application.

ARM III: Participants also receive 4 calls of 15-20 minutes each over 3 months focusing on assisting survivors with addressing challenges to receiving preventive service and health care.

ARM IV: Participants have access to EXCELS website as in Arm II. Participants also receive 4 health coaching calls as in Arm III.

Patients are followed up at 6 months, 12 months and 18 months post randomization.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with localized breast or prostate (stages 1-2) or colorectal cancer (stage 1-3)
* Have completed active treatment for their cancer diagnosis (excluding hormonal therapy)
* Have access to a phone for contact with health coach
* Be able to communicate in English; and be competent to consent
* Usability Testing and the randomized control trial (RCT): have access to a computer, a smartphone or an i-Pad/tablet equivalent with internet access

Exclusion Criteria:

* Patients who are required because of their disease to see primarily oncologists for follow-up will be excluded (i.e., those diagnosed with lymph node or distant metastasis, those with a new primary cancer)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Estimated)
Dates: Start 2013-09-03 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Use of preventive services | Up to 18 months
  Preventative services will be measured using adherence to evidence based guideline care which will be computed as a percentage of the eligible guideline related services provided to each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Shawna Hudson, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis SN, O'Malley DM, Bator A, Ohman-Strickland P, Clemow L, Ferrante JM, Crabtree BF, Miller SM, Findley P, Hudson SV. Rationale and design of extended cancer education for longer term survivors (EXCELS): a randomized control trial of 'high touch' vs. 'high tech' cancer survivorship self-management tools in primary care. BMC Cancer. 2019 Apr 11;19(1):340. doi: 10.1186/s12885-019-5531-6. PMID 30971205

DOCUMENTS (1):
  • Informed Consent Form (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT03233555/ICF_000.pdf